CLINICAL TRIAL: NCT00468312
Title: Placebo-Controlled Study of Mometasone Furoate Nasal Spray (MFNS) 200 mcg QD in the Treatment of Seasonal Allergic Rhinitis
Brief Title: Placebo-Controlled Study of Mometasone Furoate Nasal Spray (MFNS) 200 mcg QD in the Treatment of Seasonal Allergic Rhinitis (Study P05106)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05106
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone Furoate Nasal Spray (MFNS) (Experimental): 200 mcg daily
  Interventions: Drug: Mometasone furoate nasal spray
- Placebo (Placebo Comparator): Two sprays in each nostril in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone furoate nasal spray — Two sprays (50 mcg/spray) in each nostril (200 mcg daily) in the morning
  Other Names: Nasonex
  Arms: Mometasone Furoate Nasal Spray (MFNS)
Drug: Placebo — Two sprays in each nostril in the morning
  Arms: Placebo

SUMMARY:
This study is designed to assess the effectiveness of mometasone furoate nasal spray (MFNS) once daily compared with placebo in subjects with seasonal allergic rhinitis (SAR) in reducing the total symptom score.

ELIGIBILITY:
Inclusion Criteria:

* Must be 12 years of age or older, of either sex and of any race.
* Must have at least a 2-year documented history of SAR which exacerbates during the study season.
* Must have a positive skin-prick test response to an appropriate seasonal allergen at Screening (Visit 1). IgE-mediated hypersensitivity to an appropriate seasonal allergen (ie, prevailing trees and/or grasses) must be documented by a positive response to the skin prick test with wheal diameter at least 3 mm larger than diluent control after 20 minutes.
* Must be clinically symptomatic at the Screening Visit.
* Must be clinically symptomatic at the Baseline Visit.
* Must be in general good health as confirmed by routine clinical and laboratory testing and ECG results. Clinical laboratory test (CBC, blood chemistries, and urinalysis) must be within normal limits or clinically acceptable to the investigator and the sponsor.
* Must be free of any clinically significant disease, other than SAR, that would interfere with the study evaluations.
* A subject and/or a parent/guardian must be willing to give written informed consent and must be able to adhere to dosing and visit schedules and meet study requirements.
* A female subject of childbearing potential must have a negative serum pregnancy test (HCG) at Screening. Nonsterile and premenopausal female subjects must be using a medically acceptable method of birth control, ie, double barrier method, oral contraceptive, hormonal implant, or depot injectable prior to Screening and during the study.

Exclusion Criteria:

* A history of anaphylaxis and/or other severe local reaction(s) to skin testing.
* A subject with asthma who require chronic use of inhaled or systemic corticosteroids.
* Current or history of frequent, clinically significant sinusitis or chronic purulent postnasal drip.
* A subject with rhinitis medicamentosa.
* A history of allergies to more than two classes of medications or who are allergic to or cannot tolerate nasal sprays.
* A subject who have had an upper respiratory tract or sinus infection that required antibiotic therapy without at least a 14-day washout prior to the Screening Visit, or who have had a viral upper respiratory infection within 7 days before the Screening Visit.
* A subject who has nasal structural abnormalities, including large nasal polyps and marked septal deviations, which significantly interfere with nasal air flow.
* A subject who, in the opinion of the investigator, is dependent on nasal, oral, or ocular decongestants, nasal topical antihistamines, or nasal steroids.
* Use of any drug in an investigational protocol in the 30 days before the Screening Visit.
* A subject on immunotherapy (desensitization therapy), unless the subject is on a regular maintenance schedule prior to the Screening Visit and will stay on this schedule for the remainder of the study. A subject may not receive desensitization treatment within 24 hours before any visit.
* Pregnant or nursing females.
* Family member of the investigation study staff.
* Current evidence of clinically significant hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric, autoimmune disease, or other disease that precludes the subject's participation in the study. Particular attention should be given to exclude subjects with conditions that would currently interfere with the absorption, distribution, metabolism, or excretion of the study drug or interfere with the subject's ability to complete or reliably complete the diaries.
* Significant medical condition(s) that, in the judgment of the investigator, might interfere with the study or require treatment.
* A subject whose ability to provide informed consent is compromised.
* A subject with a history of noncompliance with medications or treatment

protocols.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2007-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

REFERENCES:
- [Result] Prenner BM, Lanier BQ, Bernstein DI, Shekar T, Teper A. Mometasone furoate nasal spray reduces the ocular symptoms of seasonal allergic rhinitis. J Allergy Clin Immunol. 2010 Jun;125(6):1247-1253.e5. doi: 10.1016/j.jaci.2010.03.004. PMID 20434199

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Furoate Nasal Spray (MFNS): MFNS 200 mcg (two sprays in each nostril) once daily in the morning. Each spray is equal to 50 mcg.
- Placebo: Two sprays in each nostril once daily
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Started | 220 | 209
Completed | 216 | 204
Not Completed | 4 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Did not meet protocol eligibility | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo | Total
Number analyzed (Participants) | 220 | 209 | 429
Age, Customized [Number; unit: participants] — One subject was 12 years of age at the time of enrollment/screening but turned 13 years of age at the time of randomization.
  participants
    6 - <12 years | 0 | 1 | 1
    12 - <18 years | 31 | 24 | 55
    18 - <65 years | 184 | 181 | 365
    >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 125 | 257
  Male | 88 | 84 | 172

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average AM Instantaneous (NOW) Total Nasal Symptom Score (TNSS) Averaged Over Days 2 to 15
Description: TNSS was defined as the sum of the following four nasal symptoms: rhinorrhea, nasal congestion/stuffiness, nasal itching, and sneezing; each symptom scored on a scale of 0 = none, 1 = mild, 2 = moderate, and 3 = severe. The best possible score on this scale is 0 and the worst possible score on this scale is 12.
Time Frame: Screening through 15 days daily
Population: All randomized participants were to be included in the analysis (intent-to-treat principle). However, participants with a missing evaluation at a given visit or time point were not included in the analysis for that evaluation. This included participants without a baseline score for a given change-from-baseline evaluation.
Measure: Least Squares Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 220 | 208
Score on a scale
  Baseline TNSS | 9.31 (1.60) | 9.31 (1.60)
  Change from Baseline in TNSS | -2.54 (1.99) | -1.66 (1.99)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Analysis of covariance (ANCOVA) extracted sources of variation due to treatment, variable specific baseline, and site

2. Primary Outcome: Change From Baseline in Average AM Instantaneous (NOW) Total Ocular Symptom Score (TOSS) Averaged Over Days 2 to 15
Description: TOSS was defined as the sum of the following three ocular symptoms: redness of eyes, itching/burning eyes, and tearing/watering eyes; each symptom scored on a scale of 0=none, 1=mild, 2=moderate, and 3=severe. The best possible score on this scale is 0 and the worst possible score on the scale is 9.
Time Frame: Screening through 15 days daily
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 220 | 208
Score on a scale
  Baseline TOSS | 6.78 (1.46) | 6.74 (1.46)
  Change from Baseline in TOSS | -1.71 (1.60) | -1.37 (1.60)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; p = 0.026, ANCOVA; Analysis of covariance (ANCOVA) extracted sources of variation due to treatment, variable specific baseline, and site

3. Secondary Outcome: Change From Baseline in AM NOW Nasal Congestion Score Averaged Over Days 2 to 15
Description: Nasal congestion was one of the symptoms measures in the TNSS and was scored on a scale of 0=none, 1=mild, 2=moderate, and 3=severe. The best possible score on this scale is 0 and the worst possible score on this scale is 3.
Time Frame: Screening through 15 days daily
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 220 | 208
Score on a scale
  Baseline Nasal Congestion Score | 2.60 (0.38) | 2.62 (0.38)
  change from Baseline in Nasal Congestion Score | -0.59 (0.53) | -0.39 (0.53)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Analysis of covariance (ANCOVA) extracted sources of variation due to treatment, variable specific baseline, and site

4. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Total Score at Endpoint (Last Post Baseline Evaluation Carried Forward)
Description: The RQLQ consisted of 28 items that fell into the following seven domains: activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional. Each of the items was scored from 0 = not troubled to 6 = extremely troubled, and the total of the seven domains was the primary focus of this quality of life evaluation. The best possible score on this scale is 0 and the worst possible score on this scale is 42. The Endpoint was the last post baseline evaluation carried forward and was Day 15 for the majority of the participants.
Time Frame: Baseline and 15 days
Population: The RQLQ tool is only validated in participants greater than or equal to 18 years of age. The analysis population included subjects who were randomized to treatment, answered the RQL questionnaire both at baseline and post baseline visits and were at least 18 years of age.
Measure: Least Squares Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 189 | 182
Score on a scale
  Baseline RQLQ Total Score | 4.27 (1.01) | 4.28 (1.01)
  Change from Baseline in RQLQ Total Score | -1.81 (1.36) | -1.08 (1.36)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Analysis of covariance (ANCOVA) extracted sources of variation due to treatment, variable specific baseline, and site

5. Secondary Outcome: Change From Baseline in AM Peak Nasal Inspiratory Flow (PNIF) Averaged Over Days 2 to 15
Description: Participants were to measure nasal airflow twice daily (in the morning prior to study drug dosing and in the evening) using their PNIF meter. The highest of 3 assessments was to be recorded in the electronic diary. The PNIF meter limits were between 30 and 370 liters/minute. Normal values range between 100 and 150 liters/minute. A positive change from Baseline correlates with improved nasal air flow.
Time Frame: Screening through 15 days daily
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: liters/minute
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Number analyzed (Participants) | 220 | 208
liters/minute
  Baseline PNIF | 93.12 (41.3) | 91.96 (41.3)
  Change from Baseline in PNIF | 16.55 (36.9) | 12.59 (36.9)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray (MFNS) vs Placebo; Test type: Superiority or Other; p = 0.269, ANCOVA; Analysis of covariance (ANCOVA) extracted sources of variation due to treatment, variable specific baseline, and site

ADVERSE EVENTS:
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/209
Other Adverse Events (participants affected / at risk) | 0/220 | 0/209

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 45 days from the time submitted to the sponsor for review. If the parties disagree on the communication, the investigator and sponsor's represnetatives will meet for the purpose of making a good faith effort to discuss and resolve any such issues or disagreement.